CLINICAL TRIAL: NCT07136584
Title: SOS for Caregiver Wellbeing: Testing the Feasibility of a Screening, Outcomes and Support (SOS) Model for Parents and Caregivers of Children With Chronic Conditions
Brief Title: SOS for Caregiver Wellbeing
Acronym: SOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Melbourne (Other); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HREC116190
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Mental Health; Depression and Burden in Caregivers; Anxiety Depression; Stress; Caregiver Anxiety; Parent of Child With Chronic Life-threatening Illness
Keywords: parent; caregiver; chronic illness; screening; mental health; anxiety; depression; stress; referral pathways
MeSH Terms: conditions — Psychological Well-Being; Depression; Chronic Disease; Anxiety Disorders | interventions — Mass Screening; Treatment Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening outcome - information resource sheet (Other): Arm Description
  * This is a single-arm prospective feasibility trial
  * Every consenting caregiver is screened with a mental health screening questionnaire - the Depression, Anxiety, and Stress Scale (DASS-21)
  * They will be provided feedback on their results
  * Regardless of the results, all participants will be provided an information resource sheet will that provides descriptions of common mental health conditions, details on how to access psychology support services and links to existing online mental health resources.
  Interventions: Other: Screening, Outcomes and Referral Pathways

INTERVENTIONS:
Other: Screening, Outcomes and Referral Pathways — All participants complete baseline screening with follow up at 3 and 6 months. A key feature of the study is that a standardised information resource sheet (to community-based services) is provided to all caregivers, regardless of their screening scores. Primary outcomes focus on implementation feasibility and acceptability, while secondary outcomes examine service uptake and longitudinal measurement of caregiver wellbeing.
  This differs from existing research by providing resources universally rather than only to those scoring above clinical thresholds. Our longitudinal follow-up addresses an evidence gap identified in our systematic review - limited published data on downstream effects on actual service uptake and mental health outcomes over time. The services in the resource sheet also link to routine clinical care that doesn't require specialist support programs with dedicated funding.

SUMMARY:
Parents and caregivers of children who have a chronic condition carry a large care burden and are at higher risk of having mental health symptoms. This study aims to see if completion of a mental health questionnaire by parents / caregivers at or before the child's paediatric appointment can help identify any symptoms of stress, anxiety or depression.

Following the questionnaire, parents / caregivers will be provided with the results of the questionnaire along with an information resource sheet. This will include information on anxiety, stress and depression, as well as different agencies they can contact to get support.

Parents / caregivers will be followed up at 3 and 6 months to see if they have any changes to mental health and quality of life, and whether they accessed any support services.

The primary aim for this trial is to see whether parents / caregivers find this process acceptable, and whether it can work in a busy hospital clinic.

DETAILED DESCRIPTION:
This single-arm prospective trial aims to evaluate the feasibility and acceptability of implementing a mental health screening and support pathway (the SOS model) for parents and caregivers of children with chronic conditions (CMs) in an outpatient clinic setting. The study will recruit 100 parents and caregivers attending the Royal Children's Hospital (RCH) outpatient clinics.

For the remainder of this protocol, all parents and caregivers will be referred to as 'caregivers.'

The primary objective is to test a systematic approach where:

* Caregivers undergo mental health screening using validated measures.
* Receive feedback on their mental health screening measure scores from their RCH clinician or a researcher
* All caregivers are provided with resources on appropriate support pathways

The support framework will include:

* Psychoeducational resources describing symptoms of anxiety, depression and stress
* Description of referral pathways to primary care physicians for mental health plans, enabling access to government-funded psychological support
* Connection to existing online mental health resources

By evaluating this approach, the trial seeks to determine the:

* acceptability of the screening process to both caregivers and clinicians
* feasibility of screening and feedback for caregivers attending their child's outpatient hospital appointment
* practicality of integrating mental health screening and feedback into routine outpatient care
* effectiveness of the referral pathways in connecting parents to appropriate support services
* barriers or facilitators to implementing this model of care The findings will inform whether this screening and support model could be implemented as part of standard care for caregivers of children with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* must be a parent of a child <18yo in an outpatient clinic at Royal Children's Hospital (in enrolled clinics either neuromuscular or diabetes)
* able to complete a consent form in English without an interpreter

Exclusion Criteria:

* need for an interpreter to complete informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the overall SOS Model for caregivers | Day 7
  The proportion of caregivers with a 95% confidence interval who completed screening questionnaires and received information resource sheets who report it as acceptable as measured by response to a text message: "Thinking about your recent outpatient clinic appointment with your child at The Royal Children's Hospital, did you find the SOS Model (screening, outcomes and feedback, support pathways for your own mental health and wellbeing) acceptable?" Response: Yes/No
The proportion of eligible caregivers who provide informed consent and enrol in the trial | Through study completion, an average of 6 months
  The proportion of eligible caregivers with a 95% confidence interval who provide informed consent and enrol in the trial, calculated as the number of consenting participants divided by the total number of caregivers invited to participate.
The proportion of caregivers who report following up on a recommended service on the information resource sheet on the 3-month survey. | 3 months
  The proportion of caregivers, with a 95% confidence interval, who report following up on a recommended service on the information resource sheet on the 3-month survey.
The proportion of caregivers who report following up on a recommended service on the information resource sheet on the 6-month survey. | 6 months
  The proportion of caregivers, with a 95% confidence interval, who report following up on a recommended service on the information resource sheet on the 6-month survey.

SECONDARY OUTCOMES:
The proportion of caregivers reporting comfort (acceptability) when completing the mental health survey as measured on a Likert scale on a study-designed survey | 3 months
  The proportion of caregivers, with a 95% confidence interval, who report a level of comfort when completing the mental health survey in the outpatient clinic setting using a study-designed measure in the caregiver survey Response: 5-point Likert scale ranging from 1= Very uncomfortable to 5 = Very comfortable
The proportion of caregivers who would recommend to others completing a mental health and wellbeing survey (acceptability) as measured on a Likert scale on a study-designed survey | 3 months
  The proportion of caregivers, with a 95% confidence interval, who would recommend completing a mental health and wellbeing survey to others as using a study-designed measure in the caregiver survey.
  Response: 5-point Likert scale ranging from 1= very unlikely to 5= very likely
The proportion of caregivers reporting comfort (acceptability) when discussing their survey results with a clinician as measured on a Likert scale on a study-designed survey | 3 months
  * The proportion of caregivers, with a 95% confidence interval, who report feeling comfortable discussing their mental health and wellbeing questionnaire results with one of the clinicians asked on a study-designed measure in the caregiver survey
  * Response: 5-point Likert scale ranging from 1= Very uncomfortable to 5= Very comfortable.
The proportion of clinicians who report feeling their interactions were well-received in a survey on their experience as measured on a Likert scale on a study-designed survey | 4 weeks
  The proportion of clinicians, with a 95% confidence interval, who report feeling their interactions were well-received in a survey on their experience (acceptability) Response: 5-point Likert scale ranging from 1= Not very well-received to 5= Very well-received
The proportion of clinicians who report feeling that caregivers understood the feedback results in a survey on their experience (acceptability) as measured on a Likert scale on a study-designed survey | 4 weeks
  The proportion of clinicians, with a 95% confidence interval, who report feeling that caregivers understood the feedback results in study-designed measure in a survey on their experience Response: 5-point Likert scale ranging from 1= Did not understand at all to 5= Understood very well.
The proportion of clinicians who report they found the process of discussing a caregiver's mental health easy (acceptability) in a study-designed measure in a survey on their experience | 4 weeks
  The proportion of clinicians, with a 95% confidence interval, who report they found the process of discussing a caregiver's mental health easy in a study-designed measure in a survey on their experience Response: 5-point Likert scale ranging from 1= Not easy at all to 5= Very easy
The proportion of clinicians who report they found the whole SOS model (screening, outcomes and support pathways) an acceptable addition to the clinic on a survey on their experience (acceptability) | 4 weeks
  The proportion of clinicians, with a 95% confidence interval, who report they found the whole SOS model (screening and referrals pathway) an acceptable addition to the clinic on a survey on their experience Response: Y/N
The proportion of clinicians who consent to take part in the workshop and trial (feasibility of clinician recruitment) | Through study completion, an average of 6 months
  The proportion of clinicians, with a 95% confidence interval, who take part in the workshop and trial, calculated as the number of consenting clinicians divided by the total number of caregivers invited to take part in the workshop.
The proportion of clinicians who respond that the SOS Model is feasible as per the 4-item Feasibility of Intervention Measure. | 4 weeks
  The proportion of clinicians, with a 95% confidence interval, who respond on the following Feasibility of Intervention Measure items:
  (i) The SOS Model seems implementable (ii) The SOS Model seems possible (iii) The SOS Model seems doable (iv) The SOS Model seems easy to use Response: 5-point Likert scale for each item ranging from 1 Completely disagree to 5 Completely agree
Time required for the clinician to discuss feedback and provide information as measured on a Likert scale on a study-designed survey (feasibility) | 4 weeks
  Clinicians' responses on how long on average it took to discuss feedback and provide information on a study-designed measure of their experience Response: 5-point Likert scale ranging from 1 (0-5 mins), 3 (10-15 mins) to 5 (>20 mins)
Clinician feedback on whether the mental health screening survey would add to their workload based on an open-ended question in a study designed survey (feasibility) | 4 weeks
  Study-designed, open ended question asking clinicians in what way they think this screening tool would add to their workload on a survey of their experience
The proportion of consenting caregivers who complete all study procedures | Baseline
  The proportion, with a confidence interval of 95%, of consenting caregivers who complete all procedures at baseline
The proportion of consenting caregivers who complete all study procedures | 3 months
  The proportion of consenting caregivers, with a 95% confidence interval, who complete all procedures at 3 months
The proportion of consenting caregivers who complete all study procedures | 6 months
  The proportion of consenting caregivers, with a 95% confidence interval, who complete all procedures at 6 months
The proportion of caregivers who report receiving feedback from the clinician after completing the mental health and wellbeing survey | 3 months
  The proportion of caregivers, with a 95% confidence interval, who report a clinician vs researcher provided feedback for their mental health survey. (Aiming to determine who provided the feedback).
  Response: clinician vs researcher
The proportion of caregivers who report being provided with an information resource sheet after completing their mental health and wellbeing survey (implementation fidelity) | 3 months
  The proportion of caregivers, with a 95% confidence interval, who report being provided with an information resource sheet after completing their mental health survey on a study-designed measure Response: Yes/No
The proportion of caregivers who report benefits from the referral recommendations as measured on a Likert scale on a study-designed survey | 3 months
  The proportion of caregivers, with a 95% confidence interval, who report on a study-designed survey that the recommendations on the resource sheet were useful for them Response: 5-point Likert scale ranging from 1= Not useful at all to 5= Very useful
Barriers for caregivers to take up a recommended service as measured on a multiple response question on a study-designed survey | 3 months
  The proportion of caregivers, with a 95% confidence interval, who select one or more barriers to accessing a recommendation or service as listed on a study-designed survey if they scored above the clinical cut points on the DASS-21 total score OR one or more of the subscale scores for anxiety, depression or stress
  Response:
  * I prefer to handle any problems on my own or with help from family/friends
  * I am still waiting for an appointment
  * The option was too expensive
  * It is too hard to get to
  * I do not have the time or stamina
  * The hours available for some services didn't suit
  * My health stopped me
  * Cultural or language reasons
  * I felt it would make no difference
  * I felt it would be too stressful
  * Other, please say
Changes in the mean total score between baseline and 6 months as measured on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) | Baseline, 6 months
  The comparison of mean DASS-21 total scores between baseline and 6-month follow-up among caregivers. Minimum score: 0, Maximum score: 63, Higher scores = worse outcomes.
Changes in the mean total scores of caregivers between baseline and 3 months as measured on the EuroQol five-dimensional five-level version (EQ-5D-5L) | Baseline, 3 months
  The comparison of mean EQ-5D-5L scores between baseline and 3-months follow up among caregivers. The EQ-5D-5L is a standardized instrument used to measure health-related quality of life (HRQOL). The "5D" refers to the five dimensions of health that are assessed: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The "5L" indicates that each dimension has five levels of response options, ranging from no problems to extreme problems. Scores are between 0-1.Higher scores indicate better outcomes (better health-related quality of life).
Changes in the mean total scores of caregivers between baseline and 6 months as measured on the EuroQol five-dimensional five-level version (EQ-5D-5L) | baseline, 6 months
  The comparison of mean EQ-5D-5L scores between baseline and 6-month follow up among caregivers. Scores are between 0-1. Higher scores indicate better outcomes (better health-related quality of life).
Changes in the mean total score of the visual analogue scale on the EuroQol five-dimensional five-level version (EQ-5D-5L) of caregivers between baseline and 6 months | baseline, 6 months
  The comparison in mean EQ-5D-5L visual analogue scale scores between baseline and 6-month follow up in caregivers. Scores are between 0-100. Higher scores indicate better outcomes (better self-rated health).
The proportion of caregivers with mental health scores above the cut-off scores for the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at baseline | Baseline
  The proportion of caregivers, with a 95% confidence interval, with a total score above the cut-off point (≥40) on the DASS-21 The proportion of caregivers, with a 95% confidence interval, with a subscale score above the clinical cut points: ≥14 for depression; ≥10for anxiety, and ≥19 for stress. Scores possible for each subscale: Minimum - 0, maximum - 21. Higher levels = worse outcome.
The proportion of caregivers with mental health scores above the cut off scores on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at 3 months. | 3 months
  The proportion of caregivers, with a 95% confidence interval, with a total score above the cut-off point (≥40) on the DASS-21 The proportion of caregivers, with a 95% confidence interval, with a subscale score above the clinical cut points: ≥14 for depression; ≥10for anxiety, and ≥19 for stress. Scores possible for each subscale: Minimum - 0, maximum - 21. Higher scores = worse outcome.
The proportion of caregivers with mental health scores above clinical cut off scores on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at 6 months | 6 months
  The proportion of caregivers, with a 95% confidence interval, with a total score above the cut-off point (≥40) on the DASS-21 The proportion of caregivers, with a 95% confidence interval, with a subscale score above the clinical cut points: ≥14 for depression; ≥10for anxiety, and ≥19 for stress. Scores possible for each subscale: Minimum - 0, maximum - 21. Higher score = worse outcome.
The mean total score for caregivers on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at baseline. | Baseline
  The mean total score for caregivers on the DASS-21. Scores: Minimum: 0, Maximum: 63. Higher scores = worse outcomes.
The mean total score for caregivers on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at 3 months | 3 months
  The mean total score for caregivers on the DASS-21. Scores: Minimum: 0, Maximum: 63. Higher scores = worse outcomes.
The mean total score for caregivers on the Depression, Anxiety and Stress Scale - 21-item (DASS-21) at 6 months | 6 months
  The mean total score for caregivers on the DASS-21. Total score: Scores: Minimum: 0, Maximum: 63. Higher scores = worse outcomes.
The mean total score for caregivers at baseline as measured by the EuroQol five-dimensional five-level version (EQ-5D-5L). | baseline
  The mean total score on the EQ-5D-5L in caregivers Scores are between 0-1. Higher scores indicate better outcomes (better health-related quality of life).
The mean total score for caregivers at 3 months as measured by the EuroQol five-dimensional five-level version (EQ-5D-5L). | 3 months
  The mean total score on the EQ-5D-5L in caregivers. Scores are between 0-1. Higher scores indicate better outcomes (better health-related quality of life)
The mean total score for caregivers at 6 months as measured by the EuroQol five-dimensional five-level version (EQ-5D-5L). | 6 months
  The mean total score on the EQ-5D-5L in caregivers. Scores are between 0-1. Higher scores indicate better outcomes (better health-related quality of life).
The mean total score for caregivers at baseline as measured on the visual analogue scale on the EuroQol five-dimensional five-level version (EQ-5D-5L). | baseline
  The mean total score on the visual analogue scale on the EQ-5D-5L in caregivers Scores are between 0-100. Higher scores indicate better outcomes (better self-rated health)
The mean total score for caregivers at 3 months as measured on the visual analogue scale on the EuroQol five-dimensional five-level version (EQ-5D-5L). | 3 months
  The mean total score on the visual analogue scale on the EQ-5D-5L in caregivers Scores are between 0-100. Higher scores indicate better outcomes (better self-rated health).
Changes in the mean total score between baseline and 3 months as measured on the Depression, Anxiety and Stress Scale - 21-item (DASS-21). | baseline, 3 months
  The comparison of mean DASS-21 total scores between baseline and 3-month follow-up among caregivers. Scores: Minimum: 0, Maximum: 63. Higher scores = worse outcomes.
Changes in the mean total score of the visual analogue scale of the EuroQol five-dimensional five-level version (EQ-5D-5L) at baseline and 3 months. | baseline, 3 months
  The comparison in mean EQ-5D-5L visual analogue scale scores between baseline and 3-month follow up in caregivers. Scores are between 0-100. Higher scores indicate better outcomes (better self-rated health)
The mean total score for caregivers at 6 months as measured on the visual analogue scale on the EuroQol five-dimensional five-level version (EQ-5D-5L). | 6 months
  The mean total score on the visual analogue scale on the EQ-5D-5L in caregivers Scores are between 0-100. Higher scores indicate better outcomes (better self-rated health).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Coscini, BA, MBBS, MSc, Principal Investigator — Murdoch Children's Research Institute & University of Melbourne
Locations (1):
- Outpatient clinics - Royal Children's Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared with other researchers. The specific information that will be made available includes the study protocol, statistical analysis plan, informed consent form templates, and the final report containing de-identified participant data summarised in tables and figures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months following analysis and article publication (aim August 2028), the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Murdoch Children's Research Institute's (MCRI) conditions for access:
  * Study protocol, Participant Information and Consent Forms (PICF), surveys
  * Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices)
Access Criteria: Researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access:
  * Study protocol, PICF, surveys
  * Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices)
URL: https://metis.melbournechildrens.com/

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Coscini N, McMahon G, Schulz M, Hosking C, Mulraney M, Grobler A, Hiscock H, Giallo R. Screening parents of children with a chronic condition for mental health problems: a systematic review. Arch Dis Child. 2025 Aug 18;110(9):722-728. doi: 10.1136/archdischild-2024-328300. PMID 39978866